CLINICAL TRIAL: NCT02406157
Title: Pure Yellow (577nm) Micropulse Laser Versus 532nm Subthreshold Laser Photocoagulation for Diabetic Macular Edema:A Prospective, Randomized, Paralleled Clinical Trial
Brief Title: 577nm Micropulse Laser Versus 532nm Subthreshold Laser Photocoagulation for Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZOC-MPLD
Record Dates: First submitted 2015-03-11; First posted 2015-04-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; micropulse; laser; subthreshold

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 577-MPL (Experimental): 577nm micropulse laser photocoagulation(577MPL) treatment to the macular area of retinal thickening with a focal or grid pattern
  Interventions: Device: 577-MPL
- 532-SLP (Active Comparator): 532nm subthreshold laser photocoagulation(532-SLP) treatment to the macular area of retinal thickening with a focal or grid pattern
  Interventions: Device: 532-SLP

INTERVENTIONS:
Device: 577-MPL — Device for 577nm micropulse treatment of the diabetic macular edema with the following parameters:100 microns spot size,5% duty cycle of 0.2 seconds,power is tested on micropulse mode and then reduce power to 50% of visible
  Other Names: 577nm micropulse laser photocoagulation treatment
  Arms: 577-MPL
Device: 532-SLP — Device for 532nm subthreshold treatment of the diabetic macular edema, by decomposing a subthreshold short pulse, with 10 milliseconds, 100 microns, and power(100-1000mW) adjusted according to patient's diopter transparency and pigmentation
  Other Names: 532nm subthreshold laser photocoagulation treatment
  Arms: 532-SLP

SUMMARY:
This randomized, parallel controlled, clinical-trial aims to evaluate the therapeutic efficacy and safety of 577nm micropulse laser photocoagulation for diabetic macular edema compared with 532 subthreshold laser photocoagulation.

DETAILED DESCRIPTION:
1. To evaluate the efficacy of 577nm micropulse laser photocoagulation with grid/focal treatment for diabetic macular edema.
2. To investigate influence of 577nm micropulse laser photocoagulation on structure and function of macula compared with 532nm subthreshold laser photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Patients with diabetes mellitus type 2
* Diagnosed as diabetic retinopathy with Clinical Significant Macular Edema
* Central retinal thickness(CRT) of more than 250μm as measured by optical coherence tomography (OCT)
* ETDRS visual acuity >19 letters (Snellen equivalent of 20/400 or better)
* No macular laser coagulation or surgery or medicine therapy of macular edema within the last 6 months
* Blood glucose was controlled steadily(HbA1c≤10%)

Exclusion Criteria:

* Taking part in other clinical trial within 3 months
* Planning panretinal photocoagulation(PRP) within 3 months
* Performed cataract surgery in the last 3 months
* Accompanied with other retinal vascular disease that can lead to macular edema, for example branch retinal vein occlusion(BRVO),central retinal vein occlusion(CRVO)
* Accompanied with severe opacity of refractive media that maybe impact therapy and observation
* Accompanied with nystagmus
* Accompanied with some history that maybe interfere with result or increase the risk of patients

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change of Best Corrected Visual Acuity(BCVA) | 1 year
  Best Corrected Visual Acuity will be measured by standard Early Treatment Diabetic Retinopathy Study (ETDRS) protocol

SECONDARY OUTCOMES:
Change in 10°retinal sensitivity | 1 year
  Retinal sensitivity will be measured by microperimetry
Change of fundus autofluorescence | 1 year
  Fundus autofluorescence will be evaluated for different patterns（normal, increased, and decreased）before and after treatment
Change of Central Retinal Thickness(CRT) | 1 year
  Central Retinal Thickness will be performed by optical coherence tomography(OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Lijun Zhou, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lavinsky D, Cardillo JA, Melo LA Jr, Dare A, Farah ME, Belfort R Jr. Randomized clinical trial evaluating mETDRS versus normal or high-density micropulse photocoagulation for diabetic macular edema. Invest Ophthalmol Vis Sci. 2011 Jun 17;52(7):4314-23. doi: 10.1167/iovs.10-6828. PMID 21345996